CLINICAL TRIAL: NCT06234878
Title: Validation of REEV SENSE Biomarkers Precision for Gait Analysis in Subjects With Post-stroke Gait Impairment
Brief Title: REEV SENSE for Gait Analysis in Post-stroke Gait Impairment (SENS-AG)
Acronym: SENS-AG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: REEV LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REEV-RS-01
Record Dates: First submitted 2023-12-15; First posted 2024-01-31 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Gait Disorders, Neurologic
Keywords: Stroke; Gait analysis; Accelerometer; Gait impairment
MeSH Terms: conditions — Stroke; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Gait analysis (Experimental): Gait analysis with the investigational and the reference devices
  Interventions: Device: REEV SENSE; Device: Motion capture system

INTERVENTIONS:
Device: REEV SENSE — Gait analysis with an Inertial Measurement Unit (IMU) sensor
Device: Motion capture system — Gait analysis with reflective markers and pressure sensors

SUMMARY:
The purpose of this study is to evaluate the clinical performance of the investigational REEV SENSE gait tracker to measure gait features in subjects with post-stroke gait impairment.

REEV SENSE is intended to be used by trained healthcare professionals as a simple procedure adapted to clinical routine.

The reference method for performance comparison will be motion capture.

DETAILED DESCRIPTION:
REEV SENSE is a medical device, with pending FDA and CE certifications in class 1. It is a connected gait tracker set primarily on the leg or foot, and eventually on lower limb locations. It contains an accelerometer, a certified standard battery and motion analysis algorithms that will rapidly compute easy-to-use walking analyses accessible to healthcare professionals on a mobile app.

Standard gait biomarkers such as velocity, stride length, or stance and swing times will be computed. However, REEV has also developed a new biomarker, the knee position predictor (KPP), which will provide a more accurate quantification of each individual gait profile.

The present REEV SENSE study is the first to test subjects with a pathological context, i.e. with post-stroke ambulation deficit. Performance of REEV SENSE has already been established in healthy volunteers in comparison to the reference motion capture system, indicating good technical and metrological performance.

The study will take place at the MIT Center for Clinical and Translational Research (CCTR), a reference center with a fully equipped gait lab.

Each participating volunteer will be equipped with REEV SENSE and the reference motion capture system. The participant will be asked to walk at a comfortable self selected pace for about 15 minutes back and forth along a 10m walkway. He or she may rest at any time during the walking session. REEV SENSE and motion capture data will be recorded automatically and simultaneously during the same walking session.

ELIGIBILITY:
Inclusion Criteria:

* Post-stroke gait disorder.
* Must be able to walk independently with or without the support of a cane or rollator.
* History of stroke more than six months ago.
* Be 18 years of age or older.

Exclusion Criteria:

* Subject unable to give consent.
* Subject unable to understand the tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Walking speed measure precision | Throughout study completion (an average of 2h)
  Comparison of walking speed measured with REEV SENSE with reference method

SECONDARY OUTCOMES:
KPP (Knee Position Predictor) measure precision = precision of the predicted angle of knee sagittal flexion in the next 200ms | Throughout study completion (an average of 2h)
  Comparison of KPP measured with REEV SENSE with reference method.
Walking cadence measure precision = precision of the number of steps per minute | Throughout study completion (an average of 2h)
  Comparison of walking cadence measured with REEV SENSE with reference method
Stride length measure precision | Throughout study completion (an average of 2h)
  Comparison of stride length measured with REEV SENSE with reference method
Swing time measure precision | Throughout study completion (an average of 2h)
  Comparison of swing time measured with REEV SENSE with reference method
Stance time measure precision | Throughout study completion (an average of 2h)
  Comparison of stance time measured with REEV SENSE with reference method
Stance symmetry measure precision = precision of the % of unilateral stance time predominance (right or left) compared to total bilateral stance time (right and left) | Throughout study completion (an average of 2h)
  Comparison of stance symmetry measured with REEV SENSE with reference method
Knee flexion angle measure precision in sagittal plan | Throughout study completion (an average of 2h)
  Comparison of knee flexion measured with REEV SENSE with reference method
Ankle flexion angle measure precision in sagittal plan | Throughout study completion (an average of 2h)
  Comparison of ankle flexion angle measured with REEV SENSE with reference method

CONTACTS AND LOCATIONS:
Locations (1):
- MIT Center for Clinical and Translational Research, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No